CLINICAL TRIAL: NCT05241964
Title: A Prospective Trial of Autologous Platelet-rich Plasma Injection in Erectile Dysfunction Treatment
Brief Title: Platelet-rich Plasma(PRP) Injection in ED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202008061RIPC
Record Dates: First submitted 2021-10-06; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2021-09

CONDITIONS: Erectile Dysfunction; PRP
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP (Experimental): PRP injection
  Interventions: Biological: PRP

INTERVENTIONS:
Biological: PRP — 4~6ml autologous platelet rich plasma injection every 14±2 days for a total of 5 injections.

SUMMARY:
RPR contains rich-in growth factors and has the properties of helping tissue regeneration and nerve repair. In theory, it is possibility of curing ED.

DETAILED DESCRIPTION:
There are many reasons of erectile dysfunction(ED). If left untreated, there is a major impact on relationships, self-esteem, and overall health. RPR contains rich-in growth factors and has the properties of helping tissue regeneration and nerve repair. Its mechanism is to promote the regeneration of blood vessels in the cavernous body of the penis, increase blood circulation, and then help erection, increase penile stiffness and improve the phenomenon of premature ejaculation. The main purpose of this study is to study the safety and effectiveness of PRP injection for the treatment of ED.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Between 20 and 70 years old
* Sexual dysfunction exists for at least 6 months
* IIEF-5 score 8-2
* Sign an informed consent form

Exclusion Criteria:

* Ever radical prostatectomy or extensive pelvic surgery
* Radiation therapy to the pelvic area within 12 months before recruiting
* Cancer
* Nervous system diseases that affect erectile function
* Have any blood disease
* History of coronary artery disease

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-09-22 (Estimated); Study Completion 2022-11-29 (Estimated)

PRIMARY OUTCOMES:
International Index of Erectile Function(IIEF-5) | Change from 0 week at 4,8,12,24,48 weeks
  The possible scores for the IIEF-5 range from 5 to 25, and ED was classified into five categories based on the scores: severe (5-7), moderate (8-11), mild (12-21), and no ED (22-25).

SECONDARY OUTCOMES:
Erection Hardness Score(EHS) | Change from 0 week at 4,8,12,24,48 weeks
  EHS can be a helpful tool to evaluate ED - a man's inability to get or maintain an erection firm enough for sex. To select one of the following options:
  0 Penis does not enlarge
  1. Penis is larger, but not hard
  2. Penis is hard, but not hard enough for penetration
  3. Penis is hard enough for penetration, but not completely hard
  4. Penis is completely hard and fully rigid
Duplex - Peak systolic velocity(PSV) | 0,16 weeks
  To assess penile hemodynamics - Penile arterial blood velocity record (cm/s)
Duplex - Resistance index(RI) | 0,16 weeks
  To assess penile hemodynamics - Penile vascular resistance Index

CONTACTS AND LOCATIONS:
Overall Officials: I-Ni Chiang, MD, Principal Investigator — Taipei Veteran General hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan